CLINICAL TRIAL: NCT07329166
Title: Reducing Mobility-associated Interruption in HIV Treatment in Malawi (REMIT): Pilot Trial to Assess Acceptability and Feasibility of a Mobility-specific Intervention Package
Brief Title: Reducing Mobility-associated Interruption in HIV Treatment in Malawi
Acronym: REMIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Partners in Hope, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Marguerite Thorp, MD, MPA/ID, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K01MH138243 (NIH); K01MH138243 (NIH)
Record Dates: First submitted 2026-01-08; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: mobility; antiretroviral therapy; HIV treatment interruption; ART retention; sub-Saharan Africa; Malawi; ART interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Half of facilities will be randomized to intervention status and will receive the full package of interventions, including training on mobility-specific counseling for counsellors, access to a toll-free hotline for clients and healthcare workers, and training on multi-month dispensing for providers.
  Interventions: Behavioral: REMIT intervention package
- Control (No Intervention): Half of facilities will be randomized to control status and will administer standard of care with no additional interventions offered.

INTERVENTIONS:
Behavioral: REMIT intervention package — Intervention package includes three components:
  1. Enhanced counseling: Counselors (PIH Treatment Supporters) will be trained to provide intervention counseling on mobility topics including how to prepare for travel and options for obtaining a refill while traveling.
  2. Hotline: clients and HCWs at intervention facilities will receive information about a toll-free "hotline" staffed by a treatment supporter trained in mobility-related topics. The staffer will offer advice and coordination to support mobile clients and HCWs caring for them.
  3. Training on MMD: HCWs at intervention facilities will be trained on the benefits of MMD especially for mobile clients. The MMD prescribing guidelines will be aligned with routine care and national ART guidelines, but this additional training on the benefits of MMD and its applicability to mobility will be only offered at intervention facilities.
  Arms: Intervention

SUMMARY:
The goal of this pilot clinical trial is to assess the feasibility and acceptability of an intervention package designed to reduce mobility-associated interruptions in HIV treatment in people living with HIV in Malawi who are initiating or returning to antiretroviral treatment (ART) after interruption. The main questions it aims to answer are:

* Is the intervention acceptable to healthcare workers and ART clients?
* Is the intervention feasible in the context of Malawi's health system, and what are the major operational challenges, resource requirements, and implementation barriers?

In addition, researchers will compare HIV treatment outcomes (specifically ART retention rates) between intervention and control groups to establish a preliminary estimate of the intervention's efficacy.

Participants will complete a survey on the day of enrollment and some participants will complete an in-depth interview and/or a survey after completion of the 6-month follow-up period. Facilities assigned to the intervention group will receive the full package of interventions (training on mobility-specific counseling for counsellors, access to a toll-free hotline for clients and healthcare workers, and training on multi-month dispensing for providers), while facilities assigned to the control group will provide standard of care.

DETAILED DESCRIPTION:
RATIONALE FOR RESEARCH: While Malawi has made tremendous progress towards ending the HIV epidemic - nearly reaching UNAIDS' 95-95-95 target goals (95% of people living with HIV know their status, 95% of people living with HIV have initiated ART, and 95% of those on ART reach viral suppression) - certain sub-groups of people living with HIV continue to face challenges remaining in care. One key issue that perpetuates this cycle of interruption, re-initiation, and re-interruption is mobility, or temporary travel, which is the number one reason for interruption in treatment (IIT) across several of our recent studies. Mobile people living with HIV require additional interventions to stay in care and reduce IIT. In the REMIT study (Reducing Mobility-associated Interruption in HIV Treatment), we will pilot a package of interventions that have been co-created with ART clients, healthcare workers (HCWs), and community and national stakeholders. The REMIT intervention package will include: enhanced counselling at initiation or re-initiation; a toll-free line for mobile clients and HCWs; and trainings for HCWs on the benefits of multi-month dispensing (MMD).

Study design and rationale: We propose a cluster-randomized control trial to pilot these interventions at three facilities, comparing results with three control facilities (total n=6 facilities). This cluster-randomized design is appropriate for testing interventions that are offered to healthcare workers (specifically training on an enhanced counselling curriculum and the benefits of MMD); each intervention facility will receive the full intervention package.

Population: The study population will include ART clients (≥15 years) who are initiating or re-initiating ART >28 days after a missed appointment. We will enrol n=400 men and women attending ART clinic for their own care.

We will randomly select a subset of participants from intervention facilities for additional in-depth interviews. We will also conduct focus group discussions with healthcare workers working in the ART clinic at intervention facilities.

People living with HIV and health care providers will be included in the study. Participants will be in good health so that they are feeling well and able to participate in the study. Participants will not be excluded if they are experiencing minor illness symptoms.

We will not exclude pregnant women who are otherwise eligible for the study, because they may benefit from our interventions and our interventions pose no additional risk to pregnant women relative to the general population. We will include minors aged 15-17 if they are receiving care in the general ART clinic because they may also benefit from our interventions; their participation will require parent/guardian consent and participant assent.

Research assistants will recruit participants from facilities on ART clinic days, working with facility HCWs to identify potentially eligible participants and conducting screening, consent, eligibility, and baseline survey procedures during waiting time or after the facility visit has concluded.

Interventions: Our intervention package includes three components:

1. Enhanced counseling: at facilities supported by Partners in Hope, routine care counselling is offered to clients including those initiating and re-initiating care, and covers topics such as HIV basics, disclosure, and adherence. We will be training counselors (PIH Treatment Supporters) to provide intervention counselling on mobility topics including how to prepare for travel and options for obtaining a refill while traveling.
2. Hotline: clients and HCWs at intervention facilities will receive information about a toll-free "hotline" staffed by a treatment supporter trained in mobility-related topics. The staffer will offer advice and coordination to support mobile clients and HCWs caring for them. This hotline is not part of standard of care; however, the hotline staff will provide assistance to any caller, regardless of whether they are enrolled participants or working in an intervention facility or not.
3. Training on MMD: in an effort to increase rates of MMD offered to mobile clients, we will conduct a training for HCWs at intervention facilities on the benefits of MMD especially for mobile clients. The MMD prescribing guidelines will be aligned with routine care and national ART guidelines, but this additional training on the benefits of MMD and its applicability to mobility will be only offered at intervention facilities.

Research procedures:

Baseline survey: All enrolled participants will complete a baseline survey including modules on sociodemographic characteristics and economic indicators, ART and other health history, ART knowledge, HIV stigma and disclosure status, mobility history and patterns, and other risk factors for treatment interruption including depression and alcohol use.

Implementation data: We will collect data on the implementation of the intervention, including counselling recordings, counselling progress notes, a register of calls to the hotline and call recordings, and facility-level data on MMD.

Medical chart reviews: We will conduct medical chart reviews to determine ART retention outcomes and exposure to MMD for all enrolled participants.

Follow-up survey: For all participants with chart-review evidence of treatment interruption and a subset of matched controls, we will conduct community tracing to administer a follow-up survey including updated socioeconomic and ART risk factor characteristics, verification of chart review outcomes, satisfaction with services and interventions, adverse events, and mobility during trial.

IDIs: We will conduct in-depth interviews with a subset of participants to assess intervention acceptability.

FGDs: We will conduct focus group discussions with healthcare workers to assess intervention acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. 15 years of age or older
2. Living with HIV
3. Attending ART clinic to initiate OR re-initiate care:

   1. Initiate: initiating ART for the first time, per self-report
   2. Re-initiate: returning to care after missing a refill appointment by >28 days

Exclusion Criteria:

1. Attending ART clinic on behalf of someone else (i.e. guardian)
2. Attending ART clinic only to obtain emergency refill
3. Attending ART clinic for a routine refill without a recent >=28 days interruption in treatment
4. Transferring in to study facility without a preceding interruption in treatment of >=28 days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Acceptability of REMIT intervention package | From day of intervention launch (healthcare workers) or enrollment (clients) to 6 months after final participant is enrolled
  To assess acceptability, we will analyse qualitative data from participant IDIs and HCW FGDs. We will code data from all IDIs and FGDs in Atlas.ti using inductive and deductive codes. Coded text will be analysed using grounded theory and guided by Human Centered Design principles.
Feasibility of REMIT intervention package | From day of intervention launch (healthcare workers) or enrollment (clients) to 6 months after final participant is enrolled
  To assess feasibility, we will analyse qualitative data from participant IDIs and HCW FGDs. We will code data from all IDIs and FGDs in Atlas.ti using inductive and deductive codes. Coded text will be analysed using grounded theory and guided by Human Centered Design principles. We will also review process implementation data, such as counselling recordings (fidelity of implementation and quality of counselling), the hotline register and recordings (number of calls, fidelity of implementation, and quality of counselling), and rates of MMD (compared between control and intervention facilities to assess the effectiveness of our MMD training, a component of fidelity of implementation).

SECONDARY OUTCOMES:
Preliminary estimate of efficacy | From day of enrollment to 6 months after enrollment
  We will use medical chart reviews and follow-up tracing surveys to determine rates of interruption in treatment (IIT, defined as missing an ART refill appointment by >28 days; of note, obtaining an emergency refill at another facility within 28 days of missing the appointment at a home facility will not be considered an IIT) among all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Partners in Hope, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified data (including baseline surveys conducted at enrollment, medical chart reviews, endline surveys conducted after 6-month follow-up, and summaries of in-depth interviews and focus group discussions), will be uploaded to the NIMH Data Archive.
Time Frame: By the time of publication of primary results for a minimum of 5 years.
Access Criteria: Access managed via NIMH Data Archive.